CLINICAL TRIAL: NCT01692899
Title: Retention Rates of Adalimumab, Etanercept and Infliximab as First and Second-Line Biotherapy in Patients With Rheumatoid Arthritis in Daily Practice
Acronym: MAINTAIN
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: scientific steering committee of KOL in rheumatology (Unknown)
Responsible Party: Sponsor
Other Study IDs: NRB1800007; B1801356
Record Dates: First submitted 2012-09-21; First posted 2012-09-25 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Rheumatoid Arthritis
Keywords: Retention Rates; of Adalimumab; Etanercept and Infliximab; as First and Second-Line Biotherapy; in Patients with Rheumatoid Arthritis; in Daily Practice.; TNF inhibitors; biotherapy; retrospective study
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Etanercept: Etanercept: administered as first line biotherapy in RA during the period of the study
- Adalimumab: Adalimumab: administered as first line biotherpy in RA during the period of the study
- Infliximab: Infliximab: administered as first line biotherpy in RA during the period of the study

SUMMARY:
To compare retention rates of adalimumab, etanercept and infliximab as first-line biotherapy in rheumatoid arthritis (RA), to determine causes of discontinuation, retention-associated factors, and retention rates of possible second-line tumor necrosis factor α inhibitors (TNFi).

DETAILED DESCRIPTION:
In this retrolective, multicentric study, medical charts of RA patients starting TNFi between March 2005 and April 2009 were reviewed, with follow-up between 2 and 6 years. The retention rate was estimated using the Kaplan-Meier method. Comparison between TNFi was done after adjustment using a Cox model. Factors associated with better retention were identified by multivariate analysis. Medical charts of all patients with RA starting a first TNFα inhibitor therapy between March 1, 2005 (start of commercialization of adalimumab in France) and April 30, 2009 (allowing at least 2 years of follow-up) were systematically reviewed in detail by 2 rheumatologist investigators

ELIGIBILITY:
Inclusion Criteria:

* RA defined by the 1987 ACR criteria [18]
* first TNFα inhibitor prescribed in the previously mentioned period
* TNFα inhibitor prescribed as first-line biotherapy
* undergone at least one evaluation in the center after treatment initiation

Exclusion Criteria:

* previously received another biotherapy
* TNFα inhibitor was prescribed in an RCT
* refused to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: RA defined by the 1987 ACR criteria [18]; first TNFα inhibitor prescribed in the previously mentioned period; TNFα inhibitor prescribed as first-line biotherapy; and patients had undergone at least one evaluation in the center after treatment initiation. Patients were excluded if: they had previously received another biotherapy; the TNFα inhibitor was prescribed in an RCT; or they refused to participate.
Sampling Method: Non-Probability Sample
Enrollment: 780 (Actual)
Dates: Start 2011-06; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Compare retention rates of adalimumab, etanercept and infliximab administered as first-line biologic therapy in RA | 2 years

SECONDARY OUTCOMES:
Compare retention rates of TNFα inhibitor monoclonal antibodies (adalimumab and infliximab) and the soluble receptor (etanercept) | 4 years
Causes of discontinuing these treatments | 4 years
Determine the factors associated with better retention of the first TNFα inhibitors | 4 years
Compare retention rates of possible second-line TNFα inhibitors | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- [Derived] Frazier-Mironer A, Dougados M, Mariette X, Cantagrel A, Deschamps V, Flipo RM, Logeart I, Schaeverbeke T, Sibilia J, Le Loet X, Combe B. Retention rates of adalimumab, etanercept and infliximab as first and second-line biotherapy in patients with rheumatoid arthritis in daily practice. Joint Bone Spine. 2014 Jul;81(4):352-9. doi: 10.1016/j.jbspin.2014.02.014. Epub 2014 Apr 8. PMID 24721422
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=NRB1800007&StudyName=Retention%20Rates%20of%20Adalimumab%2C%20Etanercept%20and%20Infliximab%20as%20First%20and%20Second-Line%20Biotherapy%20in%20Patients%20with%20Rheumatoid%20Arthritis%20in%20